CLINICAL TRIAL: NCT02676076
Title: A 52 WEEK, RANDOMIZED, DOUBLE BLIND, MULTINATIONAL, MULTICENTRE, ACTIVE CONTROLLED, 2-ARM PARALLEL GROUP TRIAL COMPARING CHF 5993 100/6/12.5 µg pMDI (FIXED COMBINATION OF EXTRAFINE BECLOMETASONE DIPROPIONATE PLUS FORMOTEROL FUMARATE PLUS GLYCOPYRRONIUM BROMIDE) TO CHF 1535 100/6 µg pMDI (FIXED COMBINATION OF EXTRAFINE BECLOMETHASONE DIPROPIONATE PLUS FORMOTEROL FUMARATE) IN PATIENTS WITH ASTHMA UNCONTROLLED ON MEDIUM DOSES OF INHALED CORTICOSTEROIDS IN COMBINATION WITH LONG ACTING ß2 AGONISTS
Brief Title: TRIple in asthMA With uncontRolled pAtient on Medium streNgth of ICS + LABA
Acronym: TRIMARAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-05993AB1-03; 2015-000716-18 (EudraCT Number)
Record Dates: First submitted 2016-02-03; First posted 2016-02-08 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Asthma
Keywords: asthma, anticholinergics, triple combination
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CHF 5993 100/6/12.5 µg (Experimental): Treatment A:
  CHF 5993 100/6/12.5 µg: 2 inhalations bid Total daily dose: 400/24/50 µg BDP/FF/GB
  Interventions: Drug: CHF 5993 100/6/12.5 µg
- CHF 1535 100/6 µg (Active Comparator): Treatment B :
  CHF 1535 100/6 µg: 2 inhalations bid Total daily dose: 400/24 µg BDP/FF
  Interventions: Drug: CHF 1535 100/6 µg

INTERVENTIONS:
Drug: CHF 5993 100/6/12.5 µg
  Arms: CHF 5993 100/6/12.5 µg
Drug: CHF 1535 100/6 µg
  Arms: CHF 1535 100/6 µg

SUMMARY:
The purpose of this study is to evaluate the superiority of CHF 5993 100/6/12.5 µg pMDI (fixed combination of extrafine beclometasone dipropionate plus formoterol fumarate plus glycopyrronum bromide) versus CHF 1535 100/6 µg pMDI (fixed combination of extrafine beclometasone dipropionate plus formoterol fumarate), in terms of lung functions parameters and rate of exacerbations, as well as to assess its safety and some health economics outcomes.

ELIGIBILITY:
Inclusion Criteria:

* History of asthma ≥ 1 year and diagnosed before 40 years old
* Uncontrolled asthma with double therapy only on medium doses of Inhaled CorticoSteroid (ICS) in combination with Long-acting beta2 Agonist (LABA) with ACQ-7 (Asthma Control Questionnaire) ≥1.5
* Pre-bronchodilator FEV1 <80% of the predicted normal value
* Positive reversibility test
* At least 1 documented asthma exacerbation in the previous year

Exclusion Criteria:

* Pregnant or lactating women
* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD)
* Patients with any asthma exacerbation or respiratory tract infection in the 4 weeks prior screening
* Current or ex-smokers (>= 10 packs year)
* Any change in dose, schedule or formulation of ICS + LABA combination in the 4 weeks prior screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1153 (Actual)
Dates: Start 2016-02-17 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-05-17 (Actual)

PRIMARY OUTCOMES:
Pre-dose FEV1 (Forced Expiratory Volume in the first second) | at Week 26
Reduction of moderate and severe asthma exacerbations rate | Week 0 to Week 52

SECONDARY OUTCOMES:
Peak FEV1 (Peak of Forced Expiratory Volume in the first second) within 3 hours post-dose | at Week 26
Change from baseline in morning PEF (Peak Expiratory Flow) | Week 0 to Week 26
Reduction of severe asthma exacerbations rate | Week 0 to Week 52
  Pooled analysis of CCD-05993AB1-03 and CCD-05993AB2-02 trials

OTHER OUTCOMES:
Adverse Events and Adverse Drug reactions | Up to Week 52
Collection of Health Economics outcomes | Week 0 to Week 52
  Total use of healthcare resources and absence from work

CONTACTS AND LOCATIONS:
Overall Officials: Christian Virchow, MD, Principal Investigator — Facharzt für Innere Medizin Rostock, Germany
Locations (1):
- Chiesi Clinical Trial Site 276814, Rostock, Germany

IPD SHARING:
Plan to Share IPD: Yes
Chiesi commits to sharing with qualified scientific and medical Researchers, conducting legitimate research, Patient-level Data, Study-level Data, the Clinical Protocol and the full CSR, providing access to clinical trial information consistently with the principle of safeguarding commercially confidential information and patient privacy. Any shared Patient-level Data is anonymized to protect personally identifiable information.
  Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
Access Criteria: Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
URL: https://www.chiesi.com/en/chiesi-clinical-trial-data-request-portal/

REFERENCES:
- [Result] Virchow JC, Kuna P, Paggiaro P, Papi A, Singh D, Corre S, Zuccaro F, Vele A, Kots M, Georges G, Petruzzelli S, Canonica GW. Single inhaler extrafine triple therapy in uncontrolled asthma (TRIMARAN and TRIGGER): two double-blind, parallel-group, randomised, controlled phase 3 trials. Lancet. 2019 Nov 9;394(10210):1737-1749. doi: 10.1016/S0140-6736(19)32215-9. Epub 2019 Sep 30. PMID 31582314
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] Orlovic M, Magni T, Lukyanov V, Guerra I, Madoni A. Cost-effectiveness of single-inhaler extrafine beclometasone dipropionate/formoterol fumarate/glycopyrronium in patients with uncontrolled asthma in England. Respir Med. 2022 Sep;201:106934. doi: 10.1016/j.rmed.2022.106934. Epub 2022 Jul 19. PMID 35872377
- [Derived] Papi A, Singh D, Virchow JC, Canonica GW, Vele A, Georges G. Normalisation of airflow limitation in asthma: Post-hoc analyses of TRIMARAN and TRIGGER. Clin Transl Allergy. 2022 Apr 17;12(4):e12145. doi: 10.1002/clt2.12145. eCollection 2022 Apr. PMID 35450196
- [Derived] Singh D, Virchow JC, Canonica GW, Vele A, Kots M, Georges G, Papi A. Determinants of response to inhaled extrafine triple therapy in asthma: analyses of TRIMARAN and TRIGGER. Respir Res. 2020 Oct 29;21(1):285. doi: 10.1186/s12931-020-01558-y. PMID 33121501
- [Derived] Singh D, Virchow JC, Canonica GW, Vele A, Kots M, Georges G, Papi A. Extrafine triple therapy in patients with asthma and persistent airflow limitation. Eur Respir J. 2020 Sep 24;56(3):2000476. doi: 10.1183/13993003.00476-2020. Print 2020 Sep. No abstract available. PMID 32430414
- See also: Study Record on EU Clinical Trials Register including results. — https://www.clinicaltrialsregister.eu/ctr-search/trial/2015-000716-18/results